CLINICAL TRIAL: NCT04958538
Title: A Single-cohort, Phase II Study of Methotrexate Combined Corticosteroid in Chinese Patients With Grade III-IV Acute Graft vs. Host Disease After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: MTX and Steroid for III-IV aGVHD Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Chief of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GVHD-MTX
Record Dates: First submitted 2021-06-23; First posted 2021-07-12 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Acute Graft Versus Host Disease
Keywords: acute GVHD; MTX; Corticosteroid
MeSH Terms: interventions — Methotrexate; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MTX and corticosteroid (Experimental): Methylprednisolone 2 mg/kg/day MTX (5-10 mg/day) was given on days 1, 3, and 8, and repeated weekly until aGVHD was less than grade II
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Methylprednisolone 2 mg/kg/day MTX (5-10 mg/day) was given on days 1, 3, and 8, and repeated weekly until aGVHD was less than grade II
  Other Names: Corticosteroid

SUMMARY:
The aim of the study is to identify the efficacy and safety of methotrexate (MTX) combined corticosteroid treatment for grade III-IV acute graft-versus-host disease (aGVHD) after allogeneic hematopoietic stem cell transplantation (allo-HSCT).

DETAILED DESCRIPTION:
Allo-HSCT is an effective treatment of malignant hematopoietic diseases. However, aGVHD remains a major complication after allo-HSCT and the destruction of recipient tissues by alloantigen-activated T cells is a key event in the development of aGVHD. Corticosteroid is the standard first-line therapy for aGVHD due to their roles in suppressing T cell responses. However, the response rate of corticosteroid was approximate 50%, and the clinical outcomes of patients with corticosteroid refractory GVHD were poor. Thus far, no combination therapy had been prove to be superior to corticosteroid alone as initial therapy for aGVHD. The study hypothesis: MTX combined corticosteroid treatment could help to further ameliorate the activity of T cells and control aGVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are fully informed and sign informed consent by themselves or their guardians;
2. Patients receiving allogeneic hematopoietic stem cell transplantation;
3. Patients with acute graft-versus-host disease of grade III-IV were diagnosed after transplantation;
4. Patients with stable implantation of granulocytes and platelets.

Exclusion Criteria:

1. Patients who have received more than one transplant;
2. Patients with overlap syndrome;
3. Patients within six months after the failure of the first transplantation;
4. Patients with uncontrollable active infection;
5. Patients with recurrence of primary malignant hematopathy;
6. Patients with donor lymphocyte infusion induced graft-versus-host disease after first intervention;
7. Patients with serious respiratory diseases;
8. Patients with severe renal insufficiency;
9. Patients with serious and uncontrolled heart disease;
10. Patients with severe hepatobiliary diseases unrelated to graft-versus host disease;
11. Within one week patients who need to use more than 1mg/kg/d methylprednisolone for reasons other than graft-versus-host disease;
12. patients who have participated in other clinical trials within 1 month;
13. The researcher judges that there are other factors that are not suitable for participating

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) for GVHD treatment after treatment | 14 days
  Overall response rate is defined as the proportion of patients demonstrating a complete response or partial response without requirement for additional systemic therapies for an earlier progression, mixed response or non-response

SECONDARY OUTCOMES:
Overall response rate (ORR) at 28 days after treatment | 28 days
  Overall response rate is defined as the proportion of patients demonstrating a complete response or partial response without requirement for additional systemic therapies for an earlier progression, mixed response or non-response
relapse rate | 1 year
  Relapse rate is defined as the proportion of patients demonstrating a morphological relapse of the original malignant hematological disease
Non-relapse mortality | 1 year
  Non-relapse mortality
Overall survival | 1 year
  Overall survival
Disease free survival | 1 year
  Disease free survival
Failure free survival | 1 year
  Failure free survival
Chronic GVHD | 1 year
  number of participants with chronic GVHD at one year

OTHER OUTCOMES:
Safety data (side effect) | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.Data collection including questionnaires at individual and group visits and physician interviews at individual visits will be used to assess participants for treatment-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, Dr., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University Institute of Hematology,, Beijing, Beijing Municipality, China